CLINICAL TRIAL: NCT05100173
Title: Clinical Evaluation of Genetron IDH1 PCR Kit in Glioma Patients
Status: Completed | Type: Observational
Sponsor: Genetron Health (Industry)
Collaborators: Huashan Hospital (Other); Zhejiang University (Other); West China Hospital (Other); The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016063011100922
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2017-01

CONDITIONS: Glioma, Malignant; Glioma, Mixed
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this trail is to evaluate the performance of Genetron IDH1 PCR Kit in Glioma patients using real-time PCR method.

DETAILED DESCRIPTION:
This trial follows the principle of synchronous blinding. The enrolled cases are coded, and the enrolled samples are detected with Genetron IDH1 PCR Kit and Sanger sequencing method. The results were determined independently according to the cutoff values or interpretation requirements provided by each method. Combined with the results of clinicopathological classification, the incidence of IDH1 gene R132H mutation in different subtypes was counted to evaluate the clinical performance of the Genetron IDH1 PCR Kit.

ELIGIBILITY:
Inclusion Criteria:

1. Enroll cases in strict accordance with the requirements of the study
2. The remaining samples after routine clinical testing
3. The collection and processing of samples meet the requirements of standard laboratory operations and product instructions
4. The relevant information of the sample is complete, including sample number, gender, age, and possible clinical diagnosis information
5. Each sample must have HE staining results (hematoxylin-eosin staining)
6. Pathological examination diagnosed as glioma, other brain tumors or normal tissues
7. Number of samples: 10 pieces of each sample with a thickness of 10μm, and the tumor content is not less than 50%

Exclusion Criteria:

1. Incomplete sample information
2. Severely contaminated samples
3. Samples that do not meet the requirements of sample collection and processing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital sample
Sampling Method: Non-Probability Sample
Enrollment: 1192 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2016-09-22 (Actual); Study Completion 2016-12-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of the Genetron IDH1 PCR Kit | 3 months
  The main purpose of this study is: by evaluating the Genetron IDH1 PCR Kit to compare the results of the Sanger sequencing method, and to calculate the coincidence rate and consistency of the two methods.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The First Hospital of Jilin University, Jilin
  - Huashan Hospital of Fudan University, Shanghai
  - West China Hospital of Sichuan University, Sichuan
  - The Second Affiliated Hospital of Zhejiang University, Zhejiang

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT05100173/Prot_SAP_000.pdf